CLINICAL TRIAL: NCT03496493
Title: Perioperative Comparison of the Agreement Between a Portable Fingertip Pulse Oximeter Versus Conventional Bedside Pulse Oximeter in Adult Patients
Brief Title: COMparison of Portable Fingertip Versus Conventional Pulse OximeteRs Trial
Acronym: COMFORT
Status: Completed | Type: Observational
Sponsor: University of Cape Town (Other)
Responsible Party: Principal Investigator, Ross Hofmeyr, Associate Professor, Dept Anaesthesia & Perioperative Medicine, University of Cape Town
Other Study IDs: UCT_Anaes_201801
Record Dates: First submitted 2018-01-20; First posted 2018-04-12 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Anesthesia; Hypoxemia
Keywords: perioperative; monitoring; plethysmography; pulse oximetery
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- All patients: All patients enrolled in trial will have peripheral oxygen saturation simultaneously recorded with both study devices on non-adjacent (second and fourth) fingers of the same hand.
  Interventions: Device: All patients

INTERVENTIONS:
Device: All patients — Peripheral arterial oxygen saturation recording with both study devices
  Other Names: Nihon-Kohden Lifescope BSM 3562 patient monitor; Contec CMS50D fingertip pulse oximeter

SUMMARY:
Perioperative non-invasive measurement of a patient's peripheral arterial oxygen saturation has become an accepted standard of care endorsed by anaesthesiologists and their regulatory bodies throughout the world. Pulse oximeters are an integral item on the World Health Organisation's Surgical Safety Checklist which is performed prior to the commencement of every surgical procedure. They are also utilised by other medical professionals and patients in various scenarios. When compared to conventional bedside pulse oximeters, portable fingertip devices have the advantages of cost-effectiveness, high portability, ease of use and battery operation. A review of recent literature reveals a paucity of accuracy studies in adult patients with various comorbidities in the clinical setting. Most data has been obtained under ideal laboratory conditions utilizing healthy adult volunteers. This study aims to pragmatically investigate the performance of a portable fingertip pulse oximeter in adult patients in a hospital setting.

DETAILED DESCRIPTION:
The purpose of this prospective, quantitative study is to compare the agreement between the measured arterial oxygen saturation levels using a portable fingertip versus a conventional bedside pulse oximeter in adult surgical patients, presenting for elective and emergency surgery to Groote Schuur Hospital over a four-week period. Adult surgical patients, not meeting any exclusion criteria, who present for elective or emergency surgery will be recruited. 200 data pairs (SpO2, heart rate and skin tone) will be recorded in the perioperative period (operating rooms, recovery room and intensive care unit).

Existing monitoring devices will not be disturbed. The agreement between the two devices will be compared using a Bland-Altman plot, Microsoft Excel and SPSS software. A root mean square difference value will also be calculated from these values.

No sensitive or personal patient information will be recorded, and pulse oximetry is essential harmless. Potential cross-infection will be avoided by excluding patients with known communicable diseases or open wounds/ bodily fluids in the area to have the oximeter probes applied. The study devices will be disinfected after each use. Recruitment will not affect clinical care.

The significance of this study into the performance of portable fingertip pulse oximeters in adult surgical patients will result in the availability of cheaper devices, deemed as vital anaesthetic equipment by the WHO and various anaesthetic regulatory bodies, in lower income medical facilities. It will also give anaesthetists and other medical personal the confidence to make clinical decisions based on these highly portable devices, thereby making pulse oximeters more available in resource limited areas. It will also add further data to existing studies and help assess whether darker skin pigment affects the performance of these devices in the clinical setting, which is highly relevant in an African country like South Africa.

ELIGIBILITY:
Inclusion Criteria:

* Adult surgical patients presenting for elective or emergency surgery

Exclusion Criteria:

* Contact precautions due to high risk of transmissable infectious disease
* Significant hypotension or hypoperfusion (systolic blood pressure <80 mmHg, or hypothermia)
* Motion artefacts due to excessive patient movements
* Known presence of variant haemoglobin species (eg. carboxy- or methaemoglobin)
* Intraoperative dye use (eg. methylene blue or indocyanine green)
* Nail polish or black henna
* Tape or bandages over the fingers
* Absent/inadequate pulse oximetry tracing on existing monitor

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult surgical patients presenting for elective or emergency surgery within an academic teaching hospital. Patients will have measurements made in the perioperative period in areas where conventional monitoring of pulse oximetery occurs, such as anaesthesia preassessment areas, induction rooms, operating theatres, recovery areas, ICU and PAHCU.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2018-06-11 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Saturation measurement agreement | 1 minute
  Bland-Altman analysis of saturation measurement pairs, with a priori acceptable limits of agreement (1.96 x SD measurement differences) within 3%. This is in accordance with ISO and FDA guidelines for testing of these devices (see relevant standard).

SECONDARY OUTCOMES:
Average root mean square difference | 1 minute
  Average root mean square difference in saturation pairs between the oximeters of less than 3%
Skin tone effect | 1 minute
  Subgroup analysis of effect of skin tone (Fitzpatrick scale) on oximeter agreement (provisional on adequate recruitment across groups)
Perfusion (pulse magnitude) effect on oximeter agreement | 1 minute
  Subgroup analysis of effect of magnitude of pulse waveform signal (as an indication of finger perfusion on oximeter agreement. This will be graded qualitatively as good, poor, or absent waveform, and is provisional on adequate recruitment across groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ross Hofmeyr, FCA(SA), Principal Investigator — University of Cape Town
Locations (1):
- Groote Schuur Hospital, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Raw study data will be uploaded to an open sharing platform (www.researchgate.org or similar) after publication of the study.
Supporting Information: Study Protocol, SAP
Time Frame: Upon publication of the study, to remain available indefinitely.
Access Criteria: Open access after publication